CLINICAL TRIAL: NCT02199925
Title: A Phase IV, Single-site, Open-Label Study to Evaluate the Efficacy of High-Dose Gammaplex in Children on the Autism Spectrum
Brief Title: An Open-Label Study to Evaluate the Efficacy of High-Dose Gammaplex in Children on the Autism Spectrum
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Isaac Melamed (Industry)
Collaborators: Bio Products Laboratory (Other)
Responsible Party: Sponsor-Investigator, Isaac Melamed, Principal Investigator, IMMUNOe Research Centers
Organization: IMMUNOe Research Centers (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMXAUT01
Record Dates: First submitted 2014-07-21; First posted 2014-07-25 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-03

CONDITIONS: Autism; Autistic Disorder; Asperger's Disorder; PDD; Pervasive Developmental Disorder
Keywords: Autism; Autism spectrum; Autism children
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Child Development Disorders, Pervasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gammaplex 5% IGIV (Experimental): Gammaplex 5% IGIV administered intravenously
  Interventions: Drug: Gammaplex 5%

INTERVENTIONS:
Drug: Gammaplex 5%

SUMMARY:
If autism is the consequence of a chronic inflammatory process preventing the infant brain from forming the proper neural connections, then treatment that reduces inflammation might have a positive impact on autism. IGIV treatment has been known to suppress inflammation and has been used in the treatment of inflammatory conditions and autoimmune diseases.

DETAILED DESCRIPTION:
We have come to believe that an immature immune system with abnormal signaling and altered apoptotic pathways may result in a process of neuroinflammation with a clinical presentation of Autism Spectrum Disorder. If Autism Spectrum Disorders are the consequence of a chronic inflammatory process that prevents the infant brain from forming the proper neural connections, then treatment that reduces inflammation might have a positive impact on autism. We believe that there is a correlation between immunological abnormalities and the development of the autism.

ELIGIBILITY:
Inclusion Criteria:

* The subject is between the ages of or equal to 4 and 12 years of age, of either gender, and belonging to any ethnic group.
* The subject has a diagnosis, for a minimum of 6 months prior to screening, of either autistic disorder, Asperger disorder, or pervasive developmental disorder (PDD).
* Normal physical test results.
* Immunological lab results showing reduced levels of activated CD40L or abnormal lymphocyte stimulation, or T or B cell dysfunction (hypgammaglobulinemia, primary immunodeficiency (PIDD), or common variable immune deficiency (CVID).

Exclusion Criteria:

* A diagnosis of isolated IGA deficiency
* Allergic reactions to blood products

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-04 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to assess the efficacy of Gammaplex as an immunomodulatory therapy in autistic children with evidence of immune dysfunction. | 1 year
  The primary endpoint is disease improvement, as evidenced by standardized test measures across 3 intervals: screening for baseline measurements, visit 5, and end of study visit measurements. Primary efficacy variables will be measured using the following standardized tests
  1. Caregiver Scales (SRS, CCC-2, ABC)
  2. CGI-S and CGI - I
  3. PPVT
  4. ADOS

SECONDARY OUTCOMES:
The modulatory effect of IVIG on neuroinflammation will be assessed by laboratory measurements which we believe are indicative of immune dysregulation. | 1 year

OTHER OUTCOMES:
To improve development in autistic spectrum | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Melamed, MD, Principal Investigator — IMMUNOe International Clinical Research Centers
Locations (1):
- IMMUNOe International Research Centers, Centennial, Colorado, United States